CLINICAL TRIAL: NCT01924897
Title: An Investigation Into the Role of Cardiopulmonary Exercise Testing and Pre-operative Exercise Training in Patients Undergoing Major Surgery for Colorectal Cancer
Brief Title: Preop CPET Testing and Exercise Training in Colorectal Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of East Anglia (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 2013ONC11S
Record Dates: First submitted 2013-08-14; First posted 2013-08-19 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Colorectal Neoplasms
Keywords: CPET test; Exercise training; Prehabilitation; Exercise Test
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Training Arm (Experimental): Patients randomised to exercise training will be offered three sessions of aerobic interval exercise per week over the subsequent 4 weeks prior to their procedure. Each session will comprise 6 x 5 min repetitions at 60-80% peak VO2, with 2.5 min rest intervals. The aim will be to quickly progress patients to exercise intensities that correspond to and exceed the individual AT. Heart rate, clinical signs, blood pressure and perceived exertion will be recorded regularly throughout exercise.
  Repeat CPET testing will then take place 4 weeks from the baseline test in the exercise laboratory (on the day prior to surgery) to determine changes (if any) in AT, VO2, VE/VCO2.
  Interventions: Behavioral: Exercise training
- No Exercise Training Arm (No Intervention): The patients in the non-exercise arm of the study will not undergo any exercise intervention but will be CPET tested in the exercise laboratory at the same time points as the exercise arm patients.

INTERVENTIONS:
Behavioral: Exercise training
  Arms: Exercise Training Arm

SUMMARY:
Colorectal Surgery Preoperative Exercise Training is a study being run by the colorectal surgery team at the Norfolk and Norwich University Hospital and the University of East Anglia to look at the role of exercise before surgery to improve recovery following an operation.

Having an operation to remove part of the bowel puts physical stress on the body. We know that training can help the body cope with physical stress in the same way that an athlete trains before a competition. We hypothesise that the body may recover more quickly if it is trained prior to an operation with regular and simple exercises.

Cardiopulmonary exercise testing (CPET) is used to evaluate the function of the lungs, heart and muscles at rest and during exercise. CPET testing is often done as part of standard pre-operative assessment in many hospitals for patients before undergoing major surgery. Some studies have demonstrated that CPET can be used to predict outcomes following surgery (such as time taken till discharge, complication rates).

The study consists of two parts:

Study 1) CPET variables to predict outcomes in surgery - patients will undergo a CPET test to determine baseline fitness. Blood tests will be taken around the time of surgery to examine whether biochemical markers in the bloodstream (when used in combination with results from the CPET test) can predict outcomes and recovery following colorectal surgery. Patients will then be monitored to assess their speed of recovery and rate of complications following surgery.

This will enable us to determine which CPET variables or combination of variables are most useful in the prediction of post-operative complications following colorectal surgery.

2) The second study will consist of an exercise intervention involving several sessions of supervised exercise in a laboratory. Before and at the end the exercise training regime, CPET measurements will be taken to see if fitness has improved with exercise.

This part of of the study is to determine if it is feasible to implement a structured, supervised exercise programme for patients awaiting elective colorectal cancer surgery. The results of this study will be used to inform a larger randomised controlled trial to examine the influence of exercise on CPET variables and postoperative outcomes.

DETAILED DESCRIPTION:
The study will be conducted in two parts:

Part 1. Study to examine the ability of CPET to predict outcomes in patients undergoing colorectal surgery:

Objectives

To identify which CPET variables or combination of variables are most useful in the prediction of post-operative complications following colorectal surgery. In addition, to examine whether CPET variables can be used in combination with other scoring systems or blood tests to increase accuracy of prediction. The aim of this investigation is to develop an accurate prediction model from key clinically relevant predictor variables, including CPET variables, blood tests and risk scoring systems. Such a model could be used in clinical practice to predict pre-operative outcome and thus help risk stratify patients for post-operative surveillance or management.

Study Population

The Norfolk and Norwich University Hospital undertakes approximately 300 procedures for colorectal cancers per year. Patients scheduled for cancer surgery will be recruited to the trial.

Study Outline

Informed consent to participate in the trial will be obtained in the outpatient setting after diagnosis/scheduling of surgery through discussion with the medical team and the colorectal nurse specialists. All patients will follow a standardised peri-operative pathway devised in conjunction with the surgical and anaesthetic team.

Sample Size

A sample size of a minimum of 90 patients has been identified, based on comparable studies with other patient groups in the literature.

Predictor Variables

Supervised pre-operative CPET testing will take place in the exercise laboratory at the University of East Anglia before surgery. The test is done by pedalling on a stationary bicycle, the resistance to pedalling will gradually increase, similar to when cycling up a hill. As the subject rides the stationary bike, the amount of oxygen used, and how fast/efficiently their heart beats is calculated. Breathing will be measured through a face mask or a mouth piece and the electrical activity of the heart will be measured via sensors placed on the chest. Each CPET test takes around 30 minutes to complete. For each participant in this part of the study, only one CPET test will be done prior to surgery at a convenient time.

In addition to the standard pre-surgery blood tests that all NHS patients receive, blood will be taken to measure several key serum markers which have been associated with post-operative outcomes in patients undergoing major abdominal surgery (pro-BNP, CRP, albumin and IL-6).

Scoring systems will be applied to patient data as additional indicators of peri-operative risk - these are systems which involve calculating a measure of risk based on other co-existing illnesses the patient may have.

Data Collection

Patient notes will be reviewed on each postoperative day to identify postoperative complications according to the Post-Operative Morbidity Survey system (POMS), this is a scoring tool previously used in other studies which assesses different systems of the body to determine 'morbidity' according to defined criteria (pulmonary, infection, renal, gastrointestinal, cardiovascular, wound complications, haematological and pain. Time taken until pain relief is satisfactory, ability to eat and drink, satisfactory level of mobility/self-care and bowel function will also be recorded. Length of hospital stay and time taken until the patient is medically fit for discharge will also be recorded.

Part 2: Feasibility of a randomised prehabilitation programme in patients undergoing surgery for colorectal cancer

Objectives

To determine the feasibility of implementing a structured, supervised exercise programme for patients awaiting elective colorectal cancer surgery. The results of this study will be used to inform a larger randomised controlled trial to examine the influence of exercise on CPET variables and postoperative outcomes.

Study Population (as above)

Study Outline

Following baseline CPET testing to assess initial background fitness, patients will be randomised to one of two study arms:

1. a supervised aerobic exercise training pathway + standard treatment or
2. standard treatment without supervised exercise training

To adequately assess key feasibility outcomes, a sample size of 60 patients (30 in each arm of the study) will be used.

Patients randomised to exercise training will be offered three sessions of supervised aerobic exercise per week over the subsequent 4 weeks before their procedure to be conducted in the exercise lab at the University of East Anglia.

Each session will include a few simple freehand exercises as well as some time on the treadmill or a fixed exercise bike. The sessions will last about an hour each and will be tailored to individual fitness levels. Heart rate, clinical signs, blood pressure and perceived exertion will be recorded regularly throughout exercise. This exercise protocol is currently in use in a study of elderly patients with bladder cancer awaiting surgery and is well-tolerated.

Repeat CPET testing will then take place 4 weeks from the baseline test in the exercise laboratory (on the day prior to surgery) to determine changes (if any) in CPET variables.

The patients in the non-exercise arm of the study will not undergo any exercise intervention but will be CPET tested in the exercise laboratory at the same time points as the exercise arm patients. The data from these patients (n=30) will be used to contribute to the first part of the study (CPET variables as predictors of outcome).

All patients will be CPET tested again at 3 months post-surgery to assess how well they have returned to their baseline function following their operation. Patients will be given follow-up questionnaires at this time, and again at 6 months post-surgery to assess health-related quality of life and psychological outcomes. The questionnaires used will be: CHAMPS Physical Activity Questionnaire for older adults, The Satisfaction with Life Scale, Hospital Anxiety and Depression Scale (HADS), FACT-F and the FACT-C scale to assess disease-specific quality of life.

Data collection:

As before, patient notes will be reviewed and post-operative complications identified. In addition, this study will assess the feasibility of conducting this trial on a larger scale: to identify the number of eligible patients, recruitment rate, willingness of patients to be randomised, willingness of clinicians to participate in the trial, compliance/tolerance of the exercise regimen, and patient satisfaction with the process. In addition, the costs of undergoing CPET testing and supervised exercise training will be estimated.

An assessment of key health outcomes will also be undertaken, i.e. changes in CPET variables following exercise training, postoperative complications, length of stay, and health-related quality of life benefits, thus enabling the planning of a larger trial.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Colorectal malignancy suitable for curative resection, no metastatic disease
3. Elective procedure, ability to undergo CPET testing
4. American Society of Anaesthesiologists (ASA) physical status I-III

Exclusion Criteria:

1. Emergency surgery
2. Unable to participate due to any of the following absolute contraindications to CPET testing: acute MI in past 3 - 5 days; Unstable angina; Uncontrolled arrhythmias; Syncope; Active endocarditis; Symptomatic severe aortic stenosis; Acute PE; DVT; Uncontrolled asthma; Pulmonary oedema; Room air desaturation at rest <85%; Respiratory failure; Cognitive impairment leading to inability to cooperate
3. Distant metastases on CT
4. American Society of Anaesthesiologists (ASA) physical status IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
postoperative morbidity | First 30 days following surgery
  Patient notes will be reviewed on each postoperative day to identify incidence of postoperative complications according to the Post-Operative Morbidity Survey system (POMS), a validated 18-item scoring tool which assesses nine domains of morbidity relevant to the post-surgical patient according to precisely defined criteria (pulmonary, infection, renal, gastrointestinal, cardiovascular, wound complications, haematological and pain.

SECONDARY OUTCOMES:
post-operative stay | 30 days
  total postoperative hospital stay (days postop), (including the length of stay for those patients who are readmitted to hospital within 30 days of their surgery),
mortality | 30 days
  mortality in the first 30 days following surgery will be recorded
Admission to HDU/ITU | 30 days
  The need for transfer from ward-level care to higher level care (high dependency or intensive care) following surgery

OTHER OUTCOMES:
Feasibility outcomes for exercise training | 30 days following surgery
  The primary outcomes of this study are to assess the feasibility of conducting this trial on a larger scale: to identify the number of eligible patients, recruitment rate, willingness of patients to be randomised, willingness of clinicians to participate in the trial, compliance/tolerance of the exercise regimen, patient satisfaction with the process and attrition. In addition, the costs of undergoing CPET testing and supervised exercise training will be estimated.
  An assessment of the characteristics/variability of key health outcomes will also be undertaken, i.e. changes in CPET variables following exercise training, postoperative complications, length of stay, and health-related quality of life benefits, thus enabling identification of a suitable primary outcome measure and sample size calculation for a larger trial.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University of East Anglia, Norwich, Norfolk
  - Norfolk and Norwich University Hospital, Norwich, Norfolk